CLINICAL TRIAL: NCT04506138
Title: Camrelizumab in Combination With Neoadjuvant Chemotherapy for Resectable Thoracic Esophageal Squamous Cell Carcinoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Chenqixun, Director of Thoracic Surgery Department, Zhejiang Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZJCH-2020183-II-ESCC
Record Dates: First submitted 2020-08-05; First posted 2020-08-10 (Actual); Last update posted 2021-12-14 (Actual); Status verified 2021-12

CONDITIONS: Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — camrelizumab; Paclitaxel; Injections; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Camrelizumab plus Chemotherapy (Experimental)
  Interventions: Drug: Camrelizumab; Drug: Paclitaxel for Injection (Albumin Bound); Drug: Carboplatin

INTERVENTIONS:
Drug: Camrelizumab — Camrelizumab 200mg D1, D22
Drug: Paclitaxel for Injection (Albumin Bound) — Paclitaxel for Injection (Albumin Bound) 100mg/m^2 D1, D8, D22, D29
Drug: Carboplatin — Carboplatin AUC5 D1, D22

SUMMARY:
This study aims to evaluate the efficacy of Camrelizumab with neoadjuvant chemotherapy for resectable thoracic esophageal squamous cell carcinoma

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of thoracic Esophageal squamous cell carcinoma
* ECOG performance status 0-1
* Age 18-75 years
* Resectable disease, cT2-4aNanyM0 or cT1-3N+M0
* Life expectancy more than 6 months
* Use of an effective contraceptive for adults to prevent pregnancy

Exclusion Criteria:

* Not suitable for surgery
* Prior chemotherapy, radiotherapy and immune-oncology therapies for ESCC
* Prior esophageal, gastric, or gastro-esophageal junction surgery
* Esophageal ulcer, esophageal perforation，chest pain（≥middle level）
* Pregnant or lactating women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2020-08-11 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Pathologic complete remission (PCR) | 12 weeks
Major Pathologic Response (MPR) | 12 weeks

SECONDARY OUTCOMES:
Overall Survival (OS) | 5 years
Event Free Survival（EFS） | 5 years

OTHER OUTCOMES:
EQ-5D-3L questionnaire | 5 years
FACT-E questionnaire | 5 years
  Functional Assessment of Cancer Therapy for patients with esophageal cancer questionnaire - version 4 (FACT-E)

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No